CLINICAL TRIAL: NCT01713023
Title: Effect of Fructose and Glucose and TAS1R2 in Glucose, Triglycerides, Uremia, Oxidative Stress, Feelings Related to Food Intake of Individuals With Type 1 Diabetes
Brief Title: Fructose and Glucose and TAS1R2 in Type 1 Diabetes
Acronym: TAS1R2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Débora Lopes Souto, Ph. D. student in Nutrition Sciences at the Federal University of Rio de Janeiro, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Debora-TAS1R2; CEP-151/2011 (Other Grant/Funding Number: The study received funding by FAPERJ 17/2012)
Record Dates: First submitted 2012-10-19; First posted 2012-10-24 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; fructose; glucose; TAS1R2; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose; Water; Fructose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose solution (Experimental): Solution containing 75g of glucose diluted in 200 mL of water
  Interventions: Dietary Supplement: Glucose; Dietary Supplement: Fructose
- Fructose solution (Experimental): Solution containing 75g of fructose diluted in 200 mL of water
  Interventions: Dietary Supplement: Glucose; Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Glucose — The same described in Arm description
  Other Names: 75g of glucose diluted in 200 mL of water
Dietary Supplement: Fructose — The same described in Arm description
  Other Names: 75g of fructose diluted in 200 mL of water

SUMMARY:
* BACKGROUND: Individuals with diabetes report innate preference for sweet foods, possibly due to genetic variants. In addition, studies have shown that ingestion of fructose promotes lower postprandial blood glucose, compared to glucose. However, excessive intake may increase triglycerides, uric acid and oxidative stress, due to oxidative priority.
* AIMS: To investigate the influence of fructose and glucose and taste receptor, type 1, member 2 (TAS1R2) in glucose, triglycerides, uremia, oxidative stress, feelings related to food intake and palatability of individuals with type 1 diabetes.
* METHODS: The trial is a single-blind, two-way crossover (1-week washout) study in 30 subjects with type 1 diabetes. Blood samples were collected before and 2-hours after the participants receive 75g of fructose or 75g of glucose dissolved in 200 ml water. Capillary blood glucose were assessed at 30, 90, 120, and 180 minutes to determine glucose, and visual analogue scales for measurement of appetite sensation were assessed at 70, 120, and 190 minutes.
* PURPOSE: The research proposal adds knowledge about the TAS1R2 (Ile191Val) polymorphism and around the most suitable monosaccharide for individuals with diabetes type 1.

DETAILED DESCRIPTION:
INTRODUCTION:

Fructose is transported via the portal vein to the liver, where is rapidly taken up by hepatocytes and phosphorylated to fructose-1-phosphate independent of insulin action by the enzyme fructokinase. Thus, under normal conditions, fructose is converted mainly to glucose, glycogen, and lactate, and to a small extent also to triglycerides. However a hypertriglyceridemia has been occur during high intakes of fructose.

Large amounts of fructose, unlike glucose, may result in increased lactate, pyruvate, and uric acid level in healthy subjects and patients with uncontrolled diabetes. However, uric acid also has pro-oxidative properties. Possibly, the uric acid neutralizes oxidative damage.

Sweetness is very attractive to patients with diabetes possibly due to genetic variants. The sweet taste receptor is a heterodimer of 2 protein subunits, T1R2 (taste receptor, type 1, member 2) and taste receptor, type 1, member 3, located on human chromosome 1. T1R2 is the component specific to sweet taste perception because taste receptor, type 1, member 3 is also involved in the detection of umami when it dimerizes with taste receptor, type 1, member 1.

At moment, none study assessed TAS1R variants in individuals with type 1 diabetes.

EXPERIMENTAL DESIGN:

This is a randomized, single-blind, two-way, crossover study conducted at the Research Centre (Clementino Fraga Filho University Hospital) including 30 adults with type 1 diabetes.

All volunteers will be instruct to complete the usual dietary record, register their capillary blood glucose and to abstain from vigorous physical activity, alcohol, high-fat foods and excess caffeine for 24 days before each study day.

One day before each study day, we will call to volunteer to ask about possible events that may influence the biochemical results (such as: infections, flu, fever). If we detect some, the test will be rescheduled.

Basal insulin doses will be retained, and no bolus insulin will be allowed in the morning of the day study. The study day will be performed if the blood glucose target level is between 70 and 200 mg/dL in the morning.

All volunteers will be assessed two-way crossover in a single blind, randomized fashion, with the two studies in the same subject, 1 week apart. The study was divided into two-days (the order of which was randomized): one-day with a solution containing glucose and the other with a solution containing glucose.

The subjects were admitted to the Research Centre (Nutritional Laboratory) at approximately 7-h on the day of study to test capillary blood glucose, collect arterial venous blood sample, assessed appetite sensations. After these measurements, they will rapidly drink the test solution.

Palatability ratings of the solution will assessed immediately after. Appetite sensations and will be tested using VAS scores immediately before and 70, 130, and 180 minutes after solution.

The second arterial venous blood sample will be collected 185 minutes after solution and test capillary blood glucose before and 30, 90, 120, and 180 minutes after solution.

We excluded volunteers who not complete both tests.

TEST SOLUTION Solution will be containing 75g of glucose or the same amount of fructose diluted in 200 mL of water.These amounts were calculated considering the usual oral glucose tolerance test. In addition, at moment, no studies indicate the ability capacity of fructose in patients with type 1 diabetes, however, it has been suggested that the absorption capacity of fructose in healthy adults varies from 30g to 40g.

USUAL DIETARY ASSESSMENT Usual dietary intake will be evaluated from 3-day diet records, and 24-hour recalls will be performed in the day study. All dietary records will be analyzed using a local nutritional software.

ANTHROPOMETRIC ASSESSMENT BMI will be calculated as body weight in kilograms divided by the square of height in meters.

Waist circumference will be determined as the average of two measurements calculated to the nearest 0.1cm midway between the lower rib margin and the ilial crest after a normal expiration.

Body composition will be measured by tetrapolar bioelectrical impedance(Biodynamic Model 450).

BIOCHEMICAL ASSESSMENT All arterial venous blood sample will be collected by trained healthcare professionals with disposable materials in the Research Centre (Nutritional Laboratory) and analyzed at Clinical Analysis Laboratory (located on Federal University).

Glycosylated hemoglobin, total cholesterol, HDL, creatinine, aspartate aminotransferase, alanine aminotransferase, and creatinine will be assessed to characterize the study population. Glucose, triglycerides, uric acid, pyruvic acid, lactate, and malonaldehyde will be measured before and 180 min after ingestion of solution

Glycosylated hemoglobin will be performed by high-performance liquid chromatography. Glucose, total cholesterol, HDL and triglycerides will be measured by enzymatic colorimetric method. LDL cholesterol will be calculated by Friedewald equation. Creatinine will be assessed by kinetic colorimetric method to calculates the creatinine clearance using the Cockcroft-Gault. Pyruvic acid, aspartate aminotransferase and alanine aminotransferase will be determined by ultraviolet kinetic method. Uric acid and lactate assessed by enzyme kinetic method. Malonaldehyde wil be detected by enzyme-linked immunosorbent assay.

GENOTYPING Deoxyribonucleic acid (DNA) will be isolated from whole blood using the DNA Multi-Sample Kit (Applied Biosystems®) and samples were stored at -20 degree Celsius until amplification assays in a Research Laboratory (Laboratory of Molecular Biology, Federal University).

The Ile191Val (rs35874116) polymorphism in TAS1R2 gene will be detected by using a TaqMan allelic discrimination assay (ABI number C_55646_20; Applied Biosystems, Foster City, CA) with real-time polymerase chain reaction on an ABI 7000 Sequence Detection System (Applied Biosystems). Conditions of the polymerase chain reaction is 95 degree Celsius for 10 min and 40 cycles of 95 degree Celsius for 15 s and 60 degree Celsius for 1 min. Genotyping will be verified by using positive control subjects in each 30-well plate as well as rerunning ≥ 5% of the samples, which were 100% concordant.

APPETITE AND PALATABILITY ASSESSMENT Visual analogue scales will be used to assess hunger, satiety, fullness, prospective food consumption, and palatability of the test solution, and appetite sensations will be evaluated palatability, taste, aftertaste, smell, and visual appeal of the solutions.

Both ratings consists of a visual analogue scale is a premeasured 100-mm scale that can be used to represent symptom intensity visually. Each scale is anchored at its ends by opposing feelings descriptors. Volunteers will be asked to describe their feelings by placing a vertical mark along the line that best represents the intensity of a given feelings about the solution. The distance of this mark from the appropriate anchor is measured and then translated into a score, ranging from 0 (none or best possible) to 10 (worst possible).

DIABETES TYPE 1 MANAGEMENT The investigators only included volunteers in a basal-bolus regimen with insulin infusion pump or insulin analogs (basal: detemir or glargine; bolus: lispro, glulisine or aspart) to avoid glucose oscillations during the experiment.

All volunteers will be instructed to not modify basal insulin doses and not take the morning bolus insulin. The subjects will be admitted in the Research Centre at approximately 7-h and will be test theirs capillary blood glucose, and if the blood glucose target level is between 70 and 200 mg/dL the experiment will be performed.

Before and during the experiment, we will test the capillary blood glucose levels 5-times using Accu-Check® Active, Roche, and will be canceled in glucose ≥350 mg/dL. In this case, we will take a bolus correction insulin dosage.

STATISTICAL Statistical analyzes will be performed with statistical software and significance level of 5%.

Quantitative variables will be described as the mean and standard deviation. Mann-Whitney test will be used for between-group comparison and Wilcoxon test to compare the effects of solution in each group. Spearman's correlation coefficient and regression will also be used.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes ( ≥ three years after diagnosis)
* Adults
* Normal-weight (BMI between 18.5 e 25.0 kg/m2)
* Using basal-bolus regimen with insulin infusion pump or insulin analogs (basal: detemir or glargine; bolus: lispro, glulisine or aspart).

Exclusion Criteria:

* Smokers;
* Drinkers;
* Use of exogenous hormone (with the exception of insulin);
* Use of antibiotics, anti-inflammatories or oral antidiabetics pharmacotherapy;
* Diagnosis of nephropathy;
* Diagnosis of liver diseases;
* With other types of diabetes family history;
* Visual disturbances.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Compare the effects of fructose and glucose and TAS1R2 in postprandial metabolism of individuals with type 1 diabetes | baseline up to 3 hours each day study. Total study: 2 years
  Determine the blood glucose, triglycerides, oxidation of substrates, uremia, oxidative stress, feelings related to food intake of individuals with type 1 diabetes, before and 3-hours after ingestion of 75g of fructose or 75g of glucose.

SECONDARY OUTCOMES:
Effect of fructose or glucose on blood glucose | Baseline, and up to 3-hours after solutions
  Determine the peak plasma blood glucose before and 3-hours after ingestion of 75g of fructose or 75g of glucose.
  We also test capillary blood glucose before and 30, 90, 120, and 180 minutes after solutions.
Effect of fructose or glucose on triglycerides levels | Baseline, and up to 3-hours after solutions
  Determine the triglycerides levels before and 3-hours after ingestion of 75g of fructose or 75g of glucose.
Effect of fructose or glucose on uric acid, pyruvic acid, and lactate | Baseline, and up to 3-hours after solutions
  Determine the uric acid, pyruvic acid, and lactate levels before and 3-hours after ingestion of 75g of fructose or 75g of glucose.
Effect of fructose or glucose on oxidative stress | Baseline, and up to 3-hours after solutions
  Determine the malondialdehyde level before and 3-hours after ingestion of 75g of fructose or 75g of glucose.
Effect of two polymorphisms in the gene TAS1R2 in the sweet taste perception | only at baseline
  TAS1R2 (taste receptor, type 1, member 2 T1R2) is the component specific to sweet taste perception, and does not change during the life.
  We will determine whether Ser9Cys (dbSNP: rs9701796) and Ile191Val (dbSNP: rs35874116)variations in TAS1R2 were associated with differences the sweet taste perceptions.
Effect of fructose or glucose on blood glucose | Baseline, and up to 3-hours after solutions
  Determine the peak plasma blood glucose before and 3-hours after ingestion of 75g of fructose or 75g of glucose.
  We also test capillary blood glucose before and 30, 90, 120 and 180 minutes after solutions.
Effect of fructose or glucose on appetite and palatability | Baseline, and up 120 minutes
  Two different visual analogue scales will be used to assess hunger, satiety, fullness, prospective food consumption, palatability, taste, aftertaste, smell, and visual appeal of the solutions.
  The scales will be performed at 7, 35, 95 and 120 minutes after solutions.
Effect of fructose or glucose on glucagon levels | Baseline, and up to 3-hours after solutions
  Determine the glucagon levels before and 3-hours after ingestion of 75g of fructose or 75g of glucose
Effect of fructose or glucose on leptin levels | Baseline, and up to 3-hours after solutions
  Determine the leptin levels before and 3-hours after ingestion of 75g of fructose or 75g of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Débora L Souto, Principal Investigator — Ph. D. student in Nutrition Sciences at the Federal University of Rio de Janeiro, Brazil
Locations (1):
- University Hospital of Rio de Janeiro, Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Souto DL, Lima EDS, Dantas JR, Zajdenverg L, Rodacki M, Rosado EL. Postprandial metabolic effects of fructose and glucose in type 1 diabetes patients: a pilot randomized crossover clinical trial. Arch Endocrinol Metab. 2019 Jul 29;63(4):376-384. doi: 10.20945/2359-3997000000148. PMID 31365624
- See also: Institute of Nutrition — http://www.nutricao.ufrj.br/
- See also: Federal University — http://www.hucff.ufrj.br/